CLINICAL TRIAL: NCT06886932
Title: The Effect of Pain Neuroscience Education on Patients Undergoing Surgical Repair of Moderate-Sized Rotator Cuff Tears
Brief Title: Pain Education After Rotator Cuff Surgery
Acronym: PNE-RCS
Status: Recruiting | Type: Observational
Sponsor: Elif Dilara Durmaz (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Elif Dilara Durmaz, invenstigator, Istinye University
Organization: Istinye University (Other)
Other Study IDs: IstinyeRCT2025
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Tears; Postoperative Pain Management; Shoulder Dysfunction; Kinesiophobia (Fear of Movement); Postoperative Rehabilitation
Keywords: Pain Neuroscience Education; Postoperative Rehabilitation; Rotator Cuff Tear; Kinesiophobia; Shoulder Surgery Outcomes; Postoperative Pain Management
MeSH Terms: conditions — Rotator Cuff Injuries; Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ANE + Rehabilitation (Preoperative): Patients in this group will receive Pain Neuroscience Education (ANE) before surgery, combined with a conventional rehabilitation program. The ANE will include education on pain mechanisms, neurophysiology, and the role of the central nervous system in pain perception. The conventional rehabilitation program will consist of exercises, manual therapy, and functional training tailored to rotator cuff repair recovery.
- ANE + Conventional Rehabilitation (Postoperative): Patients in this group will receive Pain Neuroscience Education (ANBE) after surgery, combined with a conventional rehabilitation program. The ANBE will focus on reducing pain catastrophizing, anxiety, and kinesiophobia, while the rehabilitation program will include postoperative exercises, mobility training, and strength-building activities.
- Conventional Rehabilitation Only (Control Group): Patients in this group will receive only the conventional rehabilitation program without any additional Pain Neuroscience Education. The rehabilitation program will include standard postoperative exercises, mobility training, and strength-building activities, as per the clinical guidelines for rotator cuff repair recovery

SUMMARY:
Study Title: The Effect of Pain Neuroscience Education Combined with Conventional Rehabilitation on Pain Management and Functional Outcomes in Patients Undergoing Mini-Open Rotator Cuff Repair

Purpose: This study aims to investigate whether adding Pain Neuroscience Education (PNE) to a conventional rehabilitation program improves pain management, physical function, and psychosocial outcomes in patients who have undergone mini-open surgery for rotator cuff tears (RCT). The study will also compare the effects of PNE when delivered before versus after surgery.

Who Can Participate: Adults aged 40-75 who have been diagnosed with a medium-sized rotator cuff tear and are scheduled for mini-open surgical repair. Participants must meet specific health criteria and be willing to participate in the rehabilitation program.

Study Details:

Participants will be randomly assigned to one of three groups:

Group 1: Conventional rehabilitation only. Group 2: Conventional rehabilitation + PNE before surgery. Group 3: Conventional rehabilitation + PNE after surgery. PNE involves educational sessions that explain the biology of pain, how the nervous system processes pain, and strategies to reduce fear and catastrophizing related to pain.

The study will last approximately 12 weeks, with regular assessments of pain levels, physical function, and psychosocial factors (e.g., fear of movement, depression, sleep quality).

Potential Benefits:

Participants may experience reduced pain, improved shoulder function, and better overall recovery.

The study may provide valuable insights into how PNE can enhance rehabilitation outcomes for patients with rotator cuff tears.

Potential Risks:

Some participants may find the educational sessions time-consuming or mentally challenging.

There is a small risk of discomfort during physical assessments or rehabilitation exercises.

Why is this study important?:

Rotator cuff tears are a common cause of shoulder pain and disability, especially in older adults. Post-surgical pain and fear of movement can slow recovery and reduce quality of life. This study will help determine whether PNE, when combined with conventional rehabilitation, can improve recovery outcomes and provide a better understanding of how timing (before or after surgery) affects its effectiveness.

DETAILED DESCRIPTION:
Background and Rationale

Rotator cuff tears (RCT) are a leading cause of shoulder pain and disability, particularly in aging populations. The prevalence of RCT increases with age, affecting approximately 28% of individuals aged 40 and rising to 60-80% in those aged 80. Surgical repair, such as mini-open rotator cuff repair, is often required for medium to large tears or when conservative treatments fail. While surgery aims to reduce pain and restore function, postoperative recovery can be challenging due to severe pain, fear of movement (kinesiophobia), and psychosocial factors like anxiety and depression. These factors can hinder rehabilitation and delay recovery.

Pain Neuroscience Education (PNE) is an evidence-based approach that teaches patients about the biological and psychological mechanisms of pain. By helping patients understand how pain is processed by the nervous system, PNE reduces fear, catastrophizing, and negative beliefs about pain, thereby improving outcomes. While PNE has been shown to be effective in chronic pain conditions, its application in acute postoperative settings, particularly for rotator cuff repair, remains underexplored.

Study Objectives

This study aims to:

Evaluate the effectiveness of combining PNE with conventional rehabilitation in improving pain management, physical function, and psychosocial outcomes in patients undergoing mini-open rotator cuff repair.

Compare the effects of delivering PNE before surgery versus after surgery. Assess the impact of PNE on secondary outcomes, including kinesiophobia, depression, pressure pain threshold, conditioned pain modulation, sleep quality, postural alignment, and functional level.

Study Design

This is a randomized controlled trial with three parallel groups:

Group 1 (Control): Conventional rehabilitation only. Group 2 (Preoperative PNE): Conventional rehabilitation + PNE delivered before surgery.

Group 3 (Postoperative PNE): Conventional rehabilitation + PNE delivered after surgery.

Methodology

Participants: Adults aged 18-65 with a diagnosed medium-sized rotator cuff tear scheduled for mini-open surgical repair.

Intervention:

PNE: A structured educational program consisting of 2-3 sessions (45-60 minutes each) that explain the neurobiology of pain, the role of the central nervous system, and strategies to reduce pain-related fear and catastrophizing.

Conventional Rehabilitation: A standardized postoperative rehabilitation program focusing on pain management, range of motion, strength training, and functional recovery.

Outcome Measures:

Primary Outcomes: Pain intensity (measured by Visual Analog Scale), shoulder function (measured by Constant-Murley Score), and kinesiophobia (measured by Tampa Scale of Kinesiophobia).

Secondary Outcomes: Depression (measured by Beck Depression Inventory), pressure pain threshold, conditioned pain modulation, sleep quality (measured by Pittsburgh Sleep Quality Index), postural alignment, and functional level.

Timeline: Participants will be assessed at baseline (pre-surgery), immediately after PNE (if applicable), and at 6 and 12 weeks post-surgery.

Statistical Analysis

Data will be analyzed using intention-to-treat principles. Repeated-measures ANOVA will be used to compare outcomes across groups and time points. Subgroup analyses will explore the effects of PNE timing (preoperative vs. postoperative).

Significance

This study addresses a critical gap in the management of rotator cuff tears by investigating the role of PNE in enhancing postoperative recovery. If effective, PNE could be integrated into standard rehabilitation protocols to improve pain management, reduce fear of movement, and accelerate functional recovery. The study also aims to determine the optimal timing for PNE delivery, providing valuable insights for clinical practice.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

Diagnosis of a medium-sized rotator cuff tear (1-3 cm) confirmed by Magnetic Resonance Imaging (MRI) and scheduled for surgical repair Age between 40 and 75 years Sufficient Turkish language proficiency to understand and complete the informed consent form and assessment scales Mini-Mental State Examination (MMSE) score ≥ 24, indicating adequate cognitive function for study participation

Exclusion Criteria:

Corticosteroid injection received within the last 6 weeks Adhesive capsulitis, defined as loss of passive external rotation greater than 50% or 30° History of previous cervical, thoracic, or shoulder surgery Presence of cervical radiculopathy, characterized by pain and tingling radiating to the arm due to nerve root involvement Acromioclavicular joint pathology or shoulder instability causing shoulder pain Full-thickness rotator cuff tear Calcific tendinitis Systemic diseases (e.g., inflammatory arthritis, malignancy) or neurological disorders (e.g., fibromyalgia, other neurological deficits) Fracture, labral lesion, or biceps tendon injury in the affected shoulder Prior participation in a chronic pain psychological management program or presence of generalized body pain

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 40-75 years who have been diagnosed with a medium-sized rotator cuff tear (1-3 cm) confirmed by Magnetic Resonance Imaging (MRI) and are scheduled for surgical repair using the mini-open surgical technique.
  Participants must meet the following inclusion criteria:
  Ability to understand and complete the informed consent form and related assessment scales in Turkish.
  A score of 24 or higher on the Mini-Mental State Examination (MMSE) to ensure adequate cognitive function for participation.
  Patients will be excluded if they have:
  Received a corticosteroid injection within the last 6 weeks. Evidence of adhesive capsulitis (loss of passive external rotation greater than 50% or 30°).
  A history of prior cervical, thoracic, or shoulder surgery. Cervical radiculopathy, acromioclavicular pathology, shoulder instability, or a full-thickness rotator cuff tear.
  Calcific tendinitis, systemic diseases (e.g., inflammatory arthritis, malignancy), o
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Time Frame: 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  Description: Pain intensity will be measured using the Numeric Analog Scale (NAS). Patients will rate their pain on a scale from 0 (no pain) to 10 (worst pain imaginable). Pain intensity will be measured using the Numeric Rating Scale (NRS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores represent worse outcomes.
Pressure Pain Threshold (PPT) | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  PPT will be measured using a digital algometer to assess changes in pain sensitivity at the shoulder region. This measures the minimum pressure required to elicit pain.
Conditioned Pain Modulation (CPM) | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  CPM will be evaluated to assess the efficiency of the endogenous pain modulation system. This measures the body's ability to modulate pain through conditioned stimuli.

SECONDARY OUTCOMES:
Kinesiophobia (Fear of Movement) | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  Kinesiophobia will be measured using the Tampa Scale of Kinesiophobia (TSK), which assesses fear of movement and reinjury.
Sleep Quality | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), which evaluates sleep duration, disturbances, and overall sleep quality.Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI total score ranges from 0 to 21, with higher scores indicating poorer sleep quality (i.e., a worse outcome).
Depression and Anxiety | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  Depression and anxiety levels will be assessed using the Depression Anxiety Stress Scale-21 (DASS-21), which consists of 21 items with three subscales: depression, anxiety, and stress. Each item is scored on a scale from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Higher scores indicate greater levels of psychological distress (i.e., a worse outcome).
Shoulder Functionality | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  Shoulder functionality will be assessed using the Shoulder Pain and Disability Index (SPADI), which evaluates pain and disability during daily activities. The total score ranges from 0 to 130, with higher scores indicating greater shoulder disability and pain (i.e., a worse outcome).
Modified Constant-Murley Shoulder Score (MCOS) | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  Shoulder Function (Modified Constant-Murley Shoulder Score) Description: Shoulder function will be evaluated using the Modified Constant-Murley Shoulder Score (MCOS), which assesses pain, activities of daily living, range of motion, and strength. The total score ranges from 0 to 100, with lower scores indicating reduced shoulder function (i.e., a worse outcome).
Functional Impairment Test-Hand, Neck, and Shoulder (FIT-HaNSA) | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  Functional impairment in the hand, neck, and shoulder regions will be assessed using the Functional Impairment Test-Hand, Neck, and Shoulder (FIT-HaNSA). The test consists of three subtasks, each performed for a maximum of 5 minutes, with specific stopping rules applied based on fatigue or inability to continue the task. Longer task durations indicate better functional capacity (i.e., a better outcome)..

OTHER OUTCOMES:
Postural Alignment | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  Postural alignment will be assessed using FizyoPrint Mobile Application, which evaluates posture and body composition. Participants will be photographed from the front, back, and side while standing in a relaxed position. The application will generate a detailed report of postural variables.
Muscle Elastography | 2 weeks before surgery (preoperative) and 8 weeks after surgery (postoperative).
  Muscle stiffness and integrity will be evaluated using Shear Wave Elastography (SWE). SWE measures the mechanical properties of the supraspinatus tendon and muscle, with higher stiffness values indicating better tissue integrity.

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data (IPD) including demographic information, clinical assessments, and key outcome measures. The data will be made available through a secure, publicly accessible data repository after the primary study results have been published. Access to the data will be provided upon request and will require submission of a research proposal for review by an independent data access committee. Data sharing will be conducted in accordance with ethical guidelines to ensure participant confidentiality and privacy.
Supporting Information: CSR, Analytic Code
Time Frame: End Date: The date when access to the data will be closed. Typically, this could be a period after the data has been shared, such as a few years after the study completion.
Access Criteria: Access will be provided through a secure, controlled-access platform (e.g., [insert platform name, e.g., ClinicalStudyDataRequest.com]).
  Researchers will need to submit a formal request and provide a research proposal. Access will be granted after approval by an independent data access committee and once a data use agreement has been signed.